CLINICAL TRIAL: NCT01087216
Title: Interest of the Dermabrasion by Laser Erbium in the Treatment of the Vitiligo
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09-PP-08; 2010-A00021-38 (Other Grant/Funding Number: AFSSAPS)
Record Dates: First submitted 2010-03-15; First posted 2010-03-16 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2010-03

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group Laser = Arm As A (Active Comparator): Opposite side lesions that will receive only the treatment by topical steroids and UVB phototherapy
  Interventions: Device: Group Laser = Arm A
- Bras B : the control group (Placebo Comparator): patient to accept habitual treatment of corticoid
  Interventions: Drug: Bras B : The group control

INTERVENTIONS:
Device: Group Laser = Arm A — Opposite side lesions that will receive only the treatment by topical steroids and UVB phototherapy
  Arms: Group Laser = Arm As A
Drug: Bras B : The group control — patient to accept habitual treatment of corticoid Opposite side lesions that will receive only the treatment by topical steroids
  Arms: Bras B : the control group

SUMMARY:
The treatment of vitiligo remains disappointing especially in some localization such as bony prominences and extremities. The association of UVB and topical steroids has been proven to be synergistic but the results are still insufficient in those difficult to treat areas. Promising results have been shown with the combination of laser assisted dermabrasion, topical 5FU and UVB. The investigators hypothesize that the dermabrasion of vitiligo skin followed by topical steroids should potentialized the effect of UVB and be superior to topical steroids and UVB without dermabrasion.

The main objective of this study is to evaluate the usefulness of laser assisted dermabrasion combined to topical steroids and UVB phototherapy in difficult to treat areas.

Patients with symmetrical non segmental vitiligo will be included in this prospective randomized monocentrer study. The investigators calculated the number of patients needed at 25. The side that will receive the dermabrasion will be centrally randomized and the opposite side will serve as control. Then on both side class 3 topical steroids will be applied daily 3 weeks on 4 for 12 weeks. UVB phototherapy will be performed twice weekly also for 12 weeks.

The evaluation will be performed by two independent physician blinded to the treatment of standardized photos before and 1 month after the end of the treatment. The criteria of success will be at least 75% of repigmentation.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 at 85
* Not segmental Vitiligo of clinical diagnosis located on bony projections or of ends
* Two symmetrical plates of vitiligo of more than 4 cm ²

Exclusion Criteria:

* Pregnant women or breastfeeding.
* Vitiligo lesions on face and neck
* Personal history of skin cancer
* Photosensitize drugs
* Personal history of photodermatosis
* Personal history of keloids
* Concomitant treatment that could have an action on vitiligo (such as tacrolimus or pimecrolimus).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-03; Primary Completion 2010-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Lesions that will receive the treatment by dermabrasion associate to habitual treatment of topical steroids and UVB phototherapy | 4 months
  Opposite side lesions that will received only the treatment by topical steroids and UVB phototherapy

CONTACTS AND LOCATIONS:
Overall Officials: PASSERON Ph Thierry, Md, Principal Investigator — CHU de Nice - Service de Dermatologie - Hôpital de l'Archet - 151 Route de saint-antoine de ginestière 06200 Nice
Locations (1):
- CHU de Nice - 4 avenue Reine Victoria - Hôpital de Cimiez, Nice, Alpes-Maritimes, France